CLINICAL TRIAL: NCT01790919
Title: Improving Depression Outcome by Enhancing Memory for Cognitive Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Allison Harvey, Professor of Clinical Psychology, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34MH094535-01A1 (NIH); R34MH094535-01A1 (NIH)
Record Dates: First submitted 2013-02-06; First posted 2013-02-13 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Depression, Adults
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Therapy plus Cognitive Support (Experimental): Cognitive therapy for depression with cognitive support added
  Interventions: Behavioral: Cognitive therapy for depression
- Cognitive therapy (Active Comparator): Cognitive therapy for depression
  Interventions: Behavioral: Cognitive therapy for depression

INTERVENTIONS:
Behavioral: Cognitive therapy for depression — Cognitive therapy (CT) for depression. There is evidence that CT for major depressive disorder (MDD) can be as effective as antidepressant medication for the initial treatment of moderate to severe MDD. Moreover, following the withdrawal of treatment, patients treated with CT are significantly less likely to relapse than patients treated with antidepressant medication and CT is at least as effective as antidepressant medication in preventing subsequent relapse. Over 14 sessions CT aims to alter the symptomatic expression of depression and reduce risk for subsequent episodes by correcting the negative beliefs and maladaptive information processing presumed to underlie the disorder and alter the systematic tendency to misperceive reality in a pessimistic fashion.
  Cognitive support. An intervention to improve memory for the contents of therapy. Cognitive support involves a series of specific procedures that support the encoding and retrieval stages of an episodic memory.

SUMMARY:
Existing drug and talking therapies for major depressive disorder (MDD) fail to produce complete recovery. This study will determine if substantial improvements to one of the most promising therapies, cognitive therapy (CT), can be achieved by administering a carefully designed procedure to improve memory for the content of CT sessions. This is important because (a) memory deficits are common in MDD patients and (b) each CT therapy session typically covers a complex array of topics and various skills are taught.

DETAILED DESCRIPTION:
Background. Major depressive disorder (MDD) is one of the most prevalent psychiatric disorders and a leading cause of disability worldwide. Existing therapies fail to produce complete recovery. Progress toward improving outcome must include innovations that are safe, powerful, inexpensive and simple (for fast and effective dissemination). The proposed research seeks to test one such innovation. We seek to improve outcome by improving memory for the content of cognitive therapy (CT) sessions. CT is one of the most promising approaches to the treatment of MDD, yet there is room for improvement.

We believe that adding memory enhancing strategies to CT may improve MDD outcome because: (a) MDD is often characterized by memory impairment, (b) there is evidence that the memory impairment is modifiable, (c) CT typically entails the activation of emotion, (d) emotion can impair or bias memory and (e) there is evidence that memory for the content of therapy sessions is poor.

Aim. To evaluate if a strategy designed to enhance memory for the content of CT sessions improves treatment outcome for MDD. Cognitive support involves a series of specific procedures that support the encoding and retrieval stages of an episodic memory. It is hypothesized that CT+Cognitive Support, relative to CT-as-usual, will be associated with improved depression outcome at the end of treatment and 6 months after the completion of treatment.

Research Plan. A small pilot feasibility RCT will be conducted on adults with MDD (n = 48) who will be randomized to one of two groups: (a) CT+Cognitive Support (n = 24) or (b) CT-as-usual (n = 24). Outcome measures will be taken at baseline, end of treatment, and 6 months after treatment. Long-term objective. To provide the pilot data needed to prepare a larger scale intervention study focused on improving outcomes by improving memory for the content of therapy sessions. The outcomes, if positive, will have major public health implications because simple, inexpensive memory enhancing strategies can be readily included as a standard feature in all psychosocial treatments for a broad range of mental illness. Project

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of major depressive disorder (MDD), first episode, recurrent or chronic, according to DSM-IV-TR criteria
* score of 24 or above on the Inventory of Depressive Symptomatology (IDS)-Clinician and 26 or above on the IDS-Self-report
* older than 18 years of age
* if taking medications for mood, medications must be stable for the past 4 weeks
* able and willing to give informed consent

Exclusion Criteria:

* history of bipolar disorder
* history of psychosis (including schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder, or psychotic organic brain syndrome)
* current non-psychotic Axis I disorder if it constitutes the principal diagnosis and if it requires treatment other than that offered in the project (including anxiety disorders including active PTSD, somatoform disorders, dissociative disorders, or eating disorders, etc.)
* history of substance dependence in the past six months
* IQ below 80
* evidence of any medical disorder or condition that could cause depression or preclude participation in CT
* current suicide risk sufficient to preclude treatment on an outpatient basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Inventory of Depressive Symptomatology, Self Report (IDS-SR) | Change in IDS scores from pre-treatment to post-treatment (defined as within 2 weeks of completing the course of treatment, which is 14 sessions) to 6-month followup
  Primary mood outcome
Global Assessment of Functioning (GAF) | Change in GAF scores from pre-treatment to post-treatment (defined as within 2 weeks of completing the course of treatment, which is 14 sessions) to 6-month followup
  Primary impairment outcome

SECONDARY OUTCOMES:
Structured Clinical Interview for DSM-IV (SCID) | Pre-treatment; Within 2 weeks of completing the course of treatment (14 sessions); 6 month followup
  To determine the presence or absence of current DSM-IV-TR defined episodes of depression
Longitudinal Interval Follow-up Evaluation (LIFE) | Pre-treatment; within 2 weeks of completing the course of treatment (14 sessions); 6-month followup
  Time to relapse or recurrence
ACNP defined Response, Remission, Relapse, Recurrence using the IDS, SCID and LIFE | Pre-treatment; within 2 weeks of completing the course of treatment (14 sessions); 6-month followup

OTHER OUTCOMES:
Memory Support Rating Scale (MSRS). | All patients receive 14 sessions of cognitive therapy for depression. The treatment sessions are video taped. A random subset of 20% of the tapes are selected for MSRS scoring. Average MSRS scores will be compared across the 2 groups.
  This is a measure of the use of memory support by treatment providers.
Patient Recall Task. | Completed at the end of Session 7, 14 and at 6 month FU. Patient Recall Task scores will be compared across the two treatment arms and over the three assessment points.
  This is a measure of the content of treatment that patient's remember
National Adult Reading Test (NART). | This measure is taken at baseline (pre-treatment) and will be compared across the two treatment arms
  Estimate of IQ. Used to determine if IQ is a moderator of treatment.
Episodic Face Naming Task. | This measure is taken at baseline (pre-treatment) and will be compared across the two treatment arms
  Measure of declarative memory. used to determine if baseline memory is a moderator of treatment outcome.
Cognitive Therapy Rating Scale (CTRS) | CTRS coding will be conducted on randomly selected recordings of treatment sessions. Average CTRS scores will be compared across the two treatment arms
  Measure of the quality of cognitive therapy
Credibility/Expectancy Questionnaire (CEQ) | The CEQ scores, measured at the end of the first therapy session, will be compared across the two treatment arms
  A measure of treatment expectancies
Demographics form | This measure is taken at baseline (pre-treatment) and will be compared across the two treatment arms
  Assesses demographics including age, years of education and chronicity of depression that are used in moderator analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

REFERENCES:
- [Derived] Dong L, Zieve G, Gumport NB, Armstrong CC, Alvarado-Martinez CG, Martinez A, Howlett S, Fine E, Tran M, McNamara ME, Weaver C, Tuck AB, Hilmoe HE, Agnew E, Fisher K, Diaz M, Lee JY, Hollon SD, Notsu H, Harvey AG. Can integrating the Memory Support Intervention into cognitive therapy improve depression outcome? A randomized controlled trial. Behav Res Ther. 2022 Oct;157:104167. doi: 10.1016/j.brat.2022.104167. Epub 2022 Aug 6. PMID 35963181
- [Derived] Harvey AG, Dong L, Lee JY, Gumport NB, Hollon SD, Rabe-Hesketh S, Hein K, Haman K, McNamara ME, Weaver C, Martinez A, Notsu H, Zieve G, Armstrong CC. Can integrating the Memory Support Intervention into cognitive therapy improve depression outcome? Study protocol for a randomized controlled trial. Trials. 2017 Nov 14;18(1):539. doi: 10.1186/s13063-017-2276-x. PMID 29137655
- [Derived] Harvey AG, Lee J, Smith RL, Gumport NB, Hollon SD, Rabe-Hesketh S, Hein K, Dolsen EA, Haman KL, Kanady JC, Thompson MA, Abrons D. Improving outcome for mental disorders by enhancing memory for treatment. Behav Res Ther. 2016 Jun;81:35-46. doi: 10.1016/j.brat.2016.03.007. Epub 2016 Apr 2. PMID 27089159